CLINICAL TRIAL: NCT00859963
Title: Regenerex Tibial Tray Multi-Center Data Collection
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.ROWG2 (US 25)
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2020-12

CONDITIONS: Pain; Arthritis
Keywords: Press fit tibial tray
MeSH Terms: conditions — Pain; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this prospective clinical data collection is to document the performance and clinical outcomes of the Regenerex™ Tibial Tray.

DETAILED DESCRIPTION:
See Protocol

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria will be identical to the indications stated in the FDA approved labeling for the device (cleared in 510(k) K080361. These indications are stated below:

1. Painful and disabled knee joint resulting from osteoarthritis, rheumatoid arthritis, traumatic arthritis where one or more compartments are involved.
2. Correction of varus, valgus, or posttraumatic deformity.
3. Correction or revision of unsuccessful osteotomy, or arthrodesis.

Patient selection factors to be considered include:

1. Ability and willingness of the patient to follow instructions, including control of weight and activity level
2. A good nutritional state of the patient, and
3. The patient must have reached full skeletal maturity

Exclusion Criteria:

The exclusion criteria will be identical to the contraindications stated in the FDA approved labeling for the device (cleared in 510(k) K080361. These contraindications are stated below:

* Absolute contraindications include: infection, sepsis, osteomyelitis, and failure of a previous joint replacement.
* Relative contraindications include:

  1. Uncooperative patient or patient with neurologic disorders who are incapable of following directions,
  2. Osteoporosis,
  3. Metabolic disorders which may impair bone formation,
  4. Osteomalacia,
  5. Distant foci of infections which may spread to the implant site,
  6. Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram,
  7. Vascular insufficiency, muscular atrophy, neuromuscular disease,
  8. Incomplete or deficient soft tissue surrounding the knee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2009-03; Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Knee Society Score | 5 years

SECONDARY OUTCOMES:
Survivorship | 5 years/ patient

CONTACTS AND LOCATIONS:
Overall Officials: Jing Xie, PhD, Study Director — Zimmer Biomet
Locations (6):
- United States (6):
  - Stanford University, Department of Orthopedics, Stanford, California
  - Midwest Orthopedics at RUSH University, Chicago, Illinois
  - Physicians Clinic of Iowa, Cedar Rapids, Iowa
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Geisinger Health System, Danville, Pennsylvania
  - Jordan-Young Institute, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: Undecided